CLINICAL TRIAL: NCT06129474
Title: DepRescribing inapprOpriate Proton Pump InhibiTors - the DROPIT Trial: a Cluster Randomized Controlled Trial in Primary Care Setting
Brief Title: Deprescribing Inappropriate Proton Pump Inhibitors
Acronym: DROPIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Swiss National Science Foundation (Other); University of Zurich (Other); University of Basel (Other); Insel Gruppe AG, University Hospital Bern (Other); Patientenstelle Zürich (Unknown); Patientenstelle Basel (Unknown); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DROPIT Trial_v1.0
Record Dates: First submitted 2023-10-23; First posted 2023-11-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Inappropriate Prescribing; Reflux Disease; Proton Pump Inhibitors
Keywords: Deprescribing; Proton pump inhibitors
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: In this trial, adult patients with inappropriate PPI prescription will be recruited by GPs in the German speaking part of Switzerland. Based on 1:1 cluster randomization of GPs, patients will be assigned to either the control group or to the group receiving an intervention to guide deprescribing of inappropriate PPIs. The control group will receive usual care.
Masking Description: Even though this is an open label study, the investigators have measures in place to mask the participants as much as possible. Patients of both groups will receive a description of the trial, which mentions inappropriate prescription of medications but not PPI, which keeps them blinded. However, GPs and patients in the intervention group may not necessarily remain blinded, since they may be questioned about the intervention as part of the integrated process evaluation of the intervention. The control group will remain unaware of the detailed nature of the intervention. In case more than one GP from a group practice takes part in this trial, GPs are instructed to keep trial-related communication and exchanges to a minimum. Team members collecting data will remain blinded to the group allocation of the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DROPIT Intervention (Experimental): The study intervention is a patient-centred PPI deprescribing intervention aiming to guide GPs and patients through the process of safely deprescribing inappropriate PPIs.
  Interventions: Other: Proton Pump Inhibitor deprescribing tool
- Usual Care (No Intervention): The reference or control arm will receive usual care. This means that the GPs and patients in this group will conduct their clinical practice as per usual, without receiving the intervention from the study team.

INTERVENTIONS:
Other: Proton Pump Inhibitor deprescribing tool — The intervention is targeted to the Swiss Primary care practice. It involves educational material and resources to guide the safe deprescribing of inappropriate PPIs, for both general practitioners and patients.
  Arms: DROPIT Intervention

SUMMARY:
The DROPIT Trial is an interventional, open-labelled, cluster-randomized controlled trial conducted in the Swiss primary care setting. It aims to evaluate an intervention to guide the deprescribing of inappropriate proton-pump inhibitors (PPIs). Therefore, the trial investigates whether the study intervention leads to the deprescribing of inappropriate PPI prescription while ensuring noninferiority safety, in comparison to usual care. Additionally, the trail aims to investigate the intervention's impact on other clinical aspects, as well as addressing features of the implementation of the intervention and its cost-effectiveness.

DETAILED DESCRIPTION:
Background and rational:

Proton pump inhibitors (PPIs) are the most frequent treatment of gastric acid related disorders. The use of PPIs is increasing, as well as concerns about their inappropriate use. Long-term use of PPIs has been associated with adverse events (e.g., nutritional deficiencies, osteoporosis, infections). Therefore, deprescribing (stopping or reducing dose) PPIs when they are not or no longer indicated is expected to benefit the patients. While general practitioners (GPs) and patients may be reluctant to deprescribing, studies suggest that clinicians would be more comfortable with deprescribing after additional training, and that patients' acceptance increases following recommendations from their doctor. This highlights the importance of providing GPs and patients with the necessary tools for safe deprescribing. In Switzerland, there is evidence of PPI use without adequate indication or dose.

In the pilot survey conducted within the current project, which involved 48 GPs, 55% of them reported often encountering patients who were prescribed inappropriate PPIs, and 58% expressed a desire for a PPI deprescribing guideline. Optimizing PPI use in Switzerland is needed and of interest. Therefore, the investigators aim to conduct a clinical trial to evaluate an intervention to guide deprescribing of inappropriate PPIs. Additionally, alongside the trial, there will be an integrated process evaluation of the intervention, and a cost-effectiveness evaluation.

Study design:

This interventional, open-labelled, cluster-randomized controlled trial in Swiss primary care setting, aims to evaluate an intervention to guide deprescribing of inappropriate PPIs. In this trial, adult patients with inappropriate PPI prescription will be recruited by GPs in the German speaking part of Switzerland. Based on 1:1 cluster randomization of GPs, patients will be assigned to either the control group or to the group receiving an intervention to guide deprescribing of inappropriate PPIs. The control group will receive usual care. The investigators will compare the effectiveness and safety of the intervention with usual care, over a 12-month follow-up period. Alongside the trial, an integrated process evaluation of the intervention and a cost-effectiveness evaluation will be conducted.

Objectives:

The main goal of this study is to evaluate an intervention to guide deprescribing of inappropriate PPIs. Therefore, the main trial aims to investigate if the study intervention leads to the deprescribing of inappropriate PPI prescription (i.e., effectiveness of the intervention), while ensuring noninferiority safety, in comparison to usual care. Additionally, the trial aims to investigate its impact on other clinical aspects, like the number of medications used, the health-related quality of life, and additional safety endpoints.

Alongside the main trial, an integrated process evaluation of the intervention aims to evaluate the quality of the implementation, as well as GPs' and patients' acceptance and fidelity to the intervention, patient typology, and the mechanisms supporting or hindering the success of the intervention.

Also, alongside the main trial, a cost-effectiveness evaluation aims to investigate the cost implications of the

Statistical considerations:

Statistical methods for the main trial The prescribed PPI dose will be quantified using the defined daily dose (DDD). To quantify its change the investigators will 1) estimate the average PPI dose over the 12 months of follow-up using the area under the curve divided by the time under observation and, 2) calculate the relative change from baseline as one minus the ratio between the average prescription and the baseline prescription level. The difference in the change in prescribed PPI dose between the two groups will be calculated using a linear model, adjusted for the baseline dose and including a random effect for the cluster. The difference in the change in upper gastrointestinal symptoms between the two groups will be calculated from a repeated-measures linear mixed-effects model, adjusted for the baseline value and including the intervention group, the timepoint, and the interaction between group and timepoint as fixed effects. Effects of the cluster and patient will be added as random effects. Both intention-to-treat (ITT) and per-protocol analyses need to meet non-inferiority to claim success for the co-primary safety endpoint.

Statistical analyses for other endpoints Repeatedly measured continuous secondary endpoints will be analyzed using the same model as for the safety co-primary endpoint. Count endpoints will be analyzed using a generalized linear mixed model and a negative binomial distribution, including the random effect of the cluster and the time of observation as an offset. Binary endpoints assessed at the end of the follow-up period will be analysed using mixed effects logistic regression, adjusted for the time under observation and including the random effect of the cluster.

Statistical methods for the integrated process evaluation of the intervention The process evaluation will be done based on the Medical Research Council's evaluation framework for complex interventions. Adherence to deprescribing decisions will be investigated using temporal dynamics modelling. Mechanisms of impact will be investigated based on the health action process approach, an established health behaviour change theory. The qualitative part will consist of semi-structured in-depth interviews with both patients and GPs.

Statistical methods for the cost-effectiveness evaluation Health economic analysis will be performed from a Swiss statutory health insurance perspective with a primary time horizon. QALYs will be estimated as the area under the survival curve resulting from utility estimates obtained for the different assessment timepoints during the trial. Utilities will be derived from EQ- 5D-5L questionnaire responses based on published valuation algorithms. A regression-based approach to assess intervention effects will be adopted due to the clustered nature of the trial data and possibility of residual baseline imbalances. The investigators will use Generalized Structural Equation Models (GSEMs), which will allow to simultaneously estimate incremental costs and QALYs (i.e., the intervention effects on costs and QALYs in the regression models), while accounting for the clustered nature of the data.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of a participating GP.
2. Age ≥18 years old.
3. Daily PPI intake for ≥8 weeks.
4. PPI twice a day or in a dose as:

   * ≥40mg/day pantoprazole;
   * ≥40mg/day omeprazole;
   * >30mg/day lansoprazole;
   * >30mg/day dexlansoprazole;
   * >20mg/day esomeprazole;
   * >20mg/day rabeprazole.
5. Sufficient knowledge of German language to understand the trial and follow-up according to GP assessment.

Exclusion Criteria:

1. Limited life expectancy according to GP judgement (patients with terminal disease and a life expectancy < 12 months.
2. Unable to provide informed consent.
3. PPI in an appropriate dose (see Appendix Table A1) and with an established indication for long-term PPI, such as:

   * History of bleeding ulcer.
   * Peptic ulcer due to cause other than NSAID or H. Pylori.
   * Barrett's oesophagus.
   * Severe erosive reflux disease (Los Angeles grade C/D).
   * GERD with symptoms or complications (oesophageal ulcer, peptic stricture).
   * Other indications (i.e., Zollinger-Ellison-Syndrome, PPI-sensitive eosinophilic esophagitis, chronic pancreatitis with steatorrhea refractory to enzyme replacement therapy, idiopathic pulmonary fibrosis.)
4. Two or more of the following medications, or one of the following medications and one or more of the below risk factors.

Medications (any dose):

* Daily use of non-steroidal anti-inflammatory drug (NSAID) >7 days.
* Antiplatelet therapy.
* Additional antiplatelet therapy (e.g., ticagrelor or similar).
* Anticoagulant(s).
* Systemic steroid(s) >1 month.

Risk factors:

* History of gastrointestinal ulcer.
* Age ≥65 years.
* Selective serotonin reuptake inhibitor (SSRI) or serotonin and norepinephrine reuptake inhibitor (SNRI) use.
* Severe concomitant disease with increased risk of GI bleeding according to the GP's assessment (e.g., severe liver disease, neoplasia, nicotine or alcohol abuse).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness co-primary endpoint: prescribed PPI dose over 12 months follow-up (superiority endpoint). | 12 months
Safety co-primary endpoint: upper gastrointestinal symptoms (Non-inferiority endpoint) | 12 months
  Co-primary endpoints measured by the Reflux Disease Questionnaire (RDQ), considering the worst of the subscales dyspepsia and gastroesophageal reflux disease (GERD) (i.e.,regurgitation and heartburn subscales combined).

SECONDARY OUTCOMES:
Occurrence of reduction of at least 50% of the prescribed PPI dose over the follow-up time. | 12 months
Occurrence of PPI discontinuation | 12 months
  Stop in PPI prescription as indicated by the general practitioner (GP)
Occurrence of PPI sustained discontinuation | 12 months
  3 months without prescribed PPI
Occurrence of a switch to prescription for on-demand use | 12 months
Occurrence of use of alternative anti-reflux treatments | 12 months
  i.e., alginate-based compounds, anti-acids, H2-blockers
Regurgitation | 12 months
  Measured with the Reflux Disease Questionnaire (RDQ). The RDQ score ranges from 0 (not present) to 5 (severe) per symptom.
Heartburn | 12 months
  Measured with the Reflux Disease Questionnaire (RDQ). The RDQ score ranges from 0 (not present) to 5 (severe) per symptom.
Dyspepsia | 12 months
  Measured with the Reflux Disease Questionnaire (RDQ). The RDQ score ranges from 0 (not present) to 5 (severe) per symptom.
Atypical gastrointestinal symptoms | 12 months
  Symptoms measured by the Reflux Symptom Index (RSI). The RSI scales for each individual item ranges from 0 (no problem) to 5 (severe problem), with a maximum total score of 45.
Occurrence of ulcers and/or gastrointestinal bleeding | 12 months
Occurrence of potential side effects of PPI overuse during the conduct of the trial. | 12 months
  Potential side effects include vitamin B12, iron (Fe), magnesium (Mg), and sodium (Na) deficiencies, osteoporosis, small intestinal bacterial overgrowth (SIBO), anemia, fractures, nephritis, and intestinal infections (C.diff., enteritis-salmonella, campylobacter).
Quality of life (EQ-5D-5L) | 12 months
  Assessed by the European Quality of Life 5-Dimensions 5-Levels (EQ-5D-5L) questionnaire. The VAS score from this questionnaire will be analyzed in the main DROPIT paper, all other questions and the resulting score will be analyzed in the health economic paper conducted alongside the trial.
Number of all medications prescribed during the conduct of the trial | 12 months
  Measured using the Anatomical Therapeutic Chemical (ATC) code

OTHER OUTCOMES:
Serious adverse events (SAE) | 12 months
  A Serious Adverse Event (SAE) (ClinO, Art. 63) is any untoward medical occurrence that results in death or is life-threatening, requires in-patient hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or causes a congenital anomaly or birth defect. Upon a SAE, the GP makes the severity assessment of the event following the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Mortality | 12 months
Patients' satisfaction with the trial participation | 12 months
  Measured by the Study Participant Feedback Questionnaire (SPFQ), handed to at the beginning (baseline), middle (6-month) and end of trial (12-month).
Use of alternative anti-reflux treatments (medication) | 12 months
  After PPI discontinuation and after PPI sustained discontinuation
New PPI prescription | 12 months
  Addressed after PPI discontinuation and after PPI sustained discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Sven Streit, Prof. Dr. med. Dr. phil, Principal Investigator — University of Bern, Institute of Primary Health Care (BIHAM)
Locations (2):
- Switzerland (2):
  - Prof. Dr. med. Dr. phil. Sven Streit, Bern
  - University of Bern, Bern

IPD SHARING:
Plan to Share IPD: Yes
Following informed consent for data sharing, data could be shared upon request to the sponsor-investigator. The data is owned by the sponsor-investigators. In case of data sharing, a data sharing agreement between the external party and the sponsor-investigator will need to be agreed on and signed.

REFERENCES:
- [Derived] Schulthess-Lisibach AE, Luthold RV, Tombez C, Weir KR, Zangger M, Chan S, Jenal F, Roumet M, Mattmann Y, Bieri C, Aubert CE, Rodondi N, Zambrano Ramos SC, Trelle S, Neuner-Jehle S, Juillerat P, Barbier M, Inauen J, Streit S, Jungo KT, Vallejo-Yague E. DepRescribing inapprOpriate Proton Pump InhibiTors (DROPIT): study protocol of a cluster-randomised controlled trial in Swiss primary care. BMJ Open. 2025 Jan 20;15(1):e094495. doi: 10.1136/bmjopen-2024-094495. PMID 39832992